CLINICAL TRIAL: NCT03255382
Title: A Randomized, Controlled, Multicenter, Open Label Study With Blinded Assessment of the Efficacy of the Humanized Anti-IL-23p19 Risankizumab Compared to FUMADERM® in Subjects With Moderate to Severe Plaque Psoriasis Who Are Naïve to and Candidates for Systemic Therapy
Brief Title: A Study to Assess the Efficacy of Risankizumab Compared to FUMADERM® in Subjects With Moderate to Severe Plaque Psoriasis Who Are Naïve to and Candidates for Systemic Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M16-178; 2016-003718-28 (EudraCT Number)
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Psoriasis
Keywords: ABBV-0066; BI 655066; risankizumab
MeSH Terms: conditions — Psoriasis | interventions — Dimethyl Fumarate; risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risankizumab (Experimental): Participants randomized to receive open-label risankizumab 150 mg by subcutaneous injection at Weeks 0, 4, and 16.
  Interventions: Drug: risankizumab
- Fumaderm (Active Comparator): Participants randomized to receive open-label Fumaderm 30 mg administered as a tablet orally once daily from Week 0 to Week 2 and then up to 240 mg, 3 times daily from Week 3 to Week 24 if 90% Improvement in Psoriasis Area and Severity Index (PASI90) is not achieved and if tolerability allows.
  Interventions: Drug: Fumaderm

INTERVENTIONS:
Drug: Fumaderm — Fumaderm tablet administered orally
  Arms: Fumaderm
Drug: risankizumab — Risankizumab administered by subcutaneous (SC) injection
  Other Names: ABBV-066; BI 655066; SKYRIZI
  Arms: Risankizumab

SUMMARY:
The purpose of this study is to compare the efficacy and safety of subcutaneous (SC) risankizumab and oral FUMADERM provided as study medication in participants with moderate to severe plaque psoriasis who are naïve to and candidates for systemic therapy.

DETAILED DESCRIPTION:
The efficacy analysis was performed in the Intent to Treat (ITT) set which included all participants who were randomized. The safety analysis was performed in the safety set which included all participants who received at least one dose of study drug. No participants were excluded from the efficacy analysis. Three participants in the FUMADERM® group discontinued after randomization prior to receiving any study drug and were thus not included in the safety set.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of chronic plaque psoriasis for at least 6 months before the first administration of study drug. Duration since diagnosis may be reported by the participant
* Participant has stable moderate to severe plaque psoriasis (body surface area [BSA] >10, Psoriasis Area and Severity Index [PASI] >10, and Dermatology Quality of Life Index [DLQI] >10) with or without psoriatic arthritis at Baseline
* Must be naïve to and candidate for systemic therapy, as assessed by the investigator
* Participant has an inadequate response, intolerance or contraindication to topical psoriasis treatment

Exclusion Criteria:

* Participants with non-plaque forms of psoriasis
* Participant has previously received systemic therapy for psoriasis, whether biologic or non-biologic or photochemotherapy
* Active systemic infection during the last 2 weeks (exception: common cold) prior to screening.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix
* Participant has any condition or contraindication to Fumaderm that would preclude the patient's participation in the present study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (23):
- Germany (23):
  - Universitaetsklinik Heidelberg /ID# 161014, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 161035, Erlangen, Bavaria
  - Universitatsklinikum Frankfurt /ID# 161036, Frankfurt am Main, Hesse
  - Universitatsklinikum Munster /ID# 165739, Munster, Lower Saxony
  - Johannes Wesling Klin Minden /ID# 161015, Minden, North Rhine-Westphalia
  - CMS3 Company for Medical Study /ID# 161103, Selters (Westerwald), Rhineland-Palatinate
  - Univ Hosp Schleswig-Holstein /ID# 160995, Kiel, Schleswig-Holstein
  - Medizinisches Versorgungszentrum DermaKiel GmbH /ID# 161102, Kiel, Schleswig-Holstein
  - Charité Universitätsmedizin Campus Mitte /ID# 165621, Berlin
  - ISA GmbH /ID# 165619, Berlin
  - Gemeinschaftspraxis /ID# 161037, Blankenfeld-mahlow
  - Hautzentrum Niesmann Othlingha /ID# 161034, Bochum
  - Universitaetsklinikum Bonn /ID# 165618, Bonn
  - Hautklinik Klinikum Darmstadt /ID# 164940, Darmstadt
  - Universitaetklinikum Dresden /ID# 160983, Dresden
  - Univ Klinik Eppendorf Hamburg /ID# 161038, Hamburg
  - Tfs /Id# 160994, Hamburg
  - Klinik fur Dermatologie /ID# 161101, Leipzig
  - Univ Johannes Gutenberg /ID# 161104, Mainz
  - TU Uniklinik Munchen /ID# 160996, Munich
  - Universitatsklinikum Tubingen /ID# 165620, Tübingen
  - Hoffmann, Witten, DE /ID# 165622, Witten
  - Centroderm Wuppertal /ID# 165615, Wuppertal

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Intent-to-treat (ITT) analysis set included all participants enrolled in the study (N = 120). Safety analysis set included all participants enrolled in the study and who received at least 1 dose of study drug (N = 117).
Pre-assignment Details: A total of 120 participants were enrolled and included in the ITT population; 3 randomized participants discontinued prior to receiving any study drug and were excluded from the safety population.
Groups:
- Fumaderm: Participants randomized to receive open-label Fumaderm 30 mg administered as a tablet orally once daily from Week 0 to Week 2, then up to 240 mg, 3 times daily from Week 3 to Week 24 if PASI90 is not achieved and if tolerability allows.
Period: Overall Study
Arm/Group | Fumaderm | Risankizumab
Started | 60 | 60
Completed | 47 | 60
Not Completed | 13 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other | 6 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) analysis set: all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fumaderm | Risankizumab | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (12.71) | 42.0 (13.75) | 42.3 (13.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 49
  Male | 38 | 33 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 59 | 60 | 119
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 60 | 59 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 90% Improvement in Psoriasis Area and Severity Index (PASI90) at Week 24
Description: The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. Non-responder imputation (NRI) was used for missing data.
Time Frame: Week 24
Population: Intent to Treat (ITT) analysis set: all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 10.0 | 83.3
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the Cochran-Mantel-Haenszel (CMH) test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 73.3, 95% CI 2-sided [61.3 to 85.3]

2. Secondary Outcome: Percentage of Participants Achieving 50% Improvement in PASI Score (PASI50) at Week 4
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI50 is defined as at least a 50% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 4
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 6.7 | 53.3
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 46.8, 95% CI 2-sided [32.8 to 60.8]

3. Secondary Outcome: Percentage of Participants Achieving 50% Improvement in PASI Score (PASI50) at Week 8
Description: as for outcome 2
Time Frame: Week 8
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 28.3 | 91.7
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 63.4, 95% CI 2-sided [50.2 to 76.6]

4. Secondary Outcome: Percentage of Participants Achieving 50% Improvement in PASI Score (PASI50) at Week 12
Description: as for outcome 2
Time Frame: Week 12
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 46.7 | 100
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 53.1, 95% CI 2-sided [40.4 to 65.7]

5. Secondary Outcome: Percentage of Participants Achieving 50% Improvement in PASI Score (PASI50) at Week 16
Description: as for outcome 2
Time Frame: Week 16
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 60.0 | 100
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 39.6, 95% CI 2-sided [27.3 to 51.9]

6. Secondary Outcome: Percentage of Participants Achieving 50% Improvement in PASI Score (PASI50) at Week 20
Description: as for outcome 2
Time Frame: Week 20
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 63.3 | 100
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 36.3, 95% CI 2-sided [24.1 to 48.5]

7. Secondary Outcome: Percentage of Participants Achieving 50% Improvement in PASI Score (PASI50) at Week 24
Description: as for outcome 2
Time Frame: Week 24
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 53.3 | 100
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 46.4, 95% CI 2-sided [33.7 to 59.0]

8. Secondary Outcome: Percentage of Participants Achieving 75% Improvement in PASI Score (PASI75) at Week 4
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI75 is defined as at least a 75% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 4
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 3.3 | 13.3
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p = 0.047, Cochran-Mantel-Haenszel; Adjusted percentage difference = 9.9, 95% CI 2-sided [0.1 to 19.7]

9. Secondary Outcome: Percentage of Participants Achieving 75% Improvement in PASI Score (PASI75) at Week 8
Description: as for outcome 8
Time Frame: Week 8
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 8.3 | 75.0
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 66.6, 95% CI 2-sided [53.8 to 79.5]

10. Secondary Outcome: Percentage of Participants Achieving 75% Improvement in PASI Score (PASI75) at Week 12
Description: as for outcome 8
Time Frame: Week 12
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 20.0 | 86.7
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 66.6, 95% CI 2-sided [53.3 to 79.9]

11. Secondary Outcome: Percentage of Participants Achieving 75% Improvement in PASI Score (PASI75) at Week 16
Description: as for outcome 8
Time Frame: Week 16
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 26.7 | 93.3
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 66.6, 95% CI 2-sided [53.8 to 79.5]

12. Secondary Outcome: Percentage of Participants Achieving 75% Improvement in PASI Score (PASI75) at Week 20
Description: as for outcome 8
Time Frame: Week 20
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 38.3 | 95.0
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 56.5, 95% CI 2-sided [43.0 to 70.0]

13. Secondary Outcome: Percentage of Participants Achieving 75% Improvement in PASI Score (PASI75) at Week 24
Description: as for outcome 8
Time Frame: Week 24
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 33.3 | 98.3
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 64.8, 95% CI 2-sided [52.5 to 77.2]

14. Secondary Outcome: Percentage of Participants Achieving 90% Improvement in PASI Score (PASI90) at Week 4
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 4
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 0 | 1.7
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p = 0.392, Cochran-Mantel-Haenszel; Adjusted percentage difference = 1.7, 95% CI 2-sided [-2.1 to 5.4]

15. Secondary Outcome: Percentage of Participants Achieving 90% Improvement in PASI Score (PASI90) at Week 8
Description: as for outcome 14
Time Frame: Week 8
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 1.7 | 38.3
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 36.6, 95% CI 2-sided [23.8 to 49.3]

16. Secondary Outcome: Percentage of Participants Achieving 90% Improvement in PASI Score (PASI90) at Week 12
Description: as for outcome 14
Time Frame: Week 12
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 5.0 | 61.7
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 56.6, 95% CI 2-sided [43.2 to 70.0]

17. Secondary Outcome: Percentage of Participants Achieving 90% Improvement in PASI Score (PASI90) at Week 16
Description: as for outcome 14
Time Frame: Week 16
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 11.7 | 76.7
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 64.9, 95% CI 2-sided [51.5 to 78.3]

18. Secondary Outcome: Percentage of Participants Achieving 90% Improvement in PASI Score (PASI90) at Week 20
Description: as for outcome 14
Time Frame: Week 20
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 16.7 | 83.3
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 66.6, 95% CI 2-sided [53.3 to 79.8]

19. Secondary Outcome: Percentage of Participants Achieving 100% Improvement in PASI (PASI100) at Week 4
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI100 is defined as 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 4
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 0 | 0
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p = 0.991, Cochran-Mantel-Haenszel; Adjusted percentage difference = 0.0, 95% CI 2-sided [-2.0 to 2.1]

20. Secondary Outcome: Percentage of Participants Achieving 100% Improvement in PASI (PASI100) at Week 8
Description: as for outcome 19
Time Frame: Week 8
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 1.7 | 5.0
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p = 0.323, Cochran-Mantel-Haenszel; Adjusted percentage difference = 3.3, 95% CI 2-sided [-3.2 to 9.8]

21. Secondary Outcome: Percentage of Participants Achieving 100% Improvement in PASI (PASI100) at Week 12
Description: as for outcome 19
Time Frame: Week 12
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 1.7 | 23.3
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 21.5, 95% CI 2-sided [10.4 to 32.6]

22. Secondary Outcome: Percentage of Participants Achieving 100% Improvement in PASI (PASI100) at Week 16
Description: as for outcome 19
Time Frame: Week 16
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Groups:
- Risankizumab: Participants randomized to receive open-label risankizumab 150 mg subcutaneous injection at Weeks 0, 4, and 16.
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 1.7 | 35.0
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 33.1, 95% CI 2-sided [20.7 to 45.5]

23. Secondary Outcome: Percentage of Participants Achieving 100% Improvement in PASI (PASI100) at Week 20
Description: as for outcome 19
Time Frame: Week 20
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 6.7 | 48.3
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 41.3, 95% CI 2-sided [27.3 to 55.3]

24. Secondary Outcome: Percentage of Participants Achieving 100% Improvement in PASI (PASI100) at Week 24
Description: as for outcome 19
Time Frame: Week 24
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 5.0 | 50.0
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 44.7, 95% CI 2-sided [30.9 to 58.5]

25. Secondary Outcome: Psoriasis Area and Severity Index (PASI): Change From Baseline to Week 4
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. Last observation carried forward (LOCF) imputation was used for missing data.
Time Frame: Baseline, Week 4
Population: ITT analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
units on a scale | -2.37 (0.669) | -9.56 (0.673)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and the treatment in this model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -7.19, 95% CI 2-sided [-8.82 to -5.56], Standard Error of Mean 0.825

26. Secondary Outcome: PASI: Change From Baseline to Week 8
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 8
Population: ITT analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 58 | 60
units on a scale | -5.61 (0.759) | -15.18 (0.763)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -9.58, 95% CI 2-sided [-11.43 to -7.72], Standard Error of Mean 0.936

27. Secondary Outcome: PASI: Change From Baseline to Week 12
Description: as for outcome 26
Time Frame: Baseline, Week 12
Population: ITT analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 58 | 60
units on a scale | -7.69 (0.788) | -16.49 (0.793)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -8.80, 95% CI 2-sided [-10.72 to -6.87], Standard Error of Mean 0.972

28. Secondary Outcome: PASI: Change From Baseline to Week 16
Description: as for outcome 26
Time Frame: Baseline, Week 16
Population: ITT analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 58 | 60
units on a scale | -9.11 (0.777) | -16.89 (0.782)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -7.78, 95% CI 2-sided [-9.68 to -5.88], Standard Error of Mean 0.958

29. Secondary Outcome: PASI: Change From Baseline to Week 20
Description: as for outcome 26
Time Frame: Baseline, Week 20
Population: ITT analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 58 | 60
units on a scale | -9.46 (0.894) | -17.35 (0.899)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -7.89, 95% CI 2-sided [-10.07 to -5.71], Standard Error of Mean 1.101

30. Secondary Outcome: PASI: Change From Baseline to Week 24
Description: as for outcome 26
Time Frame: Baseline, Week 24
Population: ITT analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 58 | 60
units on a scale | -9.31 (0.953) | -17.69 (0.959)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -8.39, 95% CI 2-sided [-10.71 to -6.06], Standard Error of Mean 1.175

31. Secondary Outcome: Percentage of Participants Achieving Static Physician Global Assessment (sPGA) Score of Clear or Almost Clear at Week 4
Description: The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA ranges from 0 to 4, and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5. NRI was used for missing data.
Time Frame: Week 4
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 3.3 | 33.3
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 29.7, 95% CI 2-sided [17.1 to 42.4]

32. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear or Almost Clear at Week 8
Description: as for outcome 31
Time Frame: Week 8
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 15.0 | 81.7
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 66.7, 95% CI 2-sided [53.4 to 80.0]

33. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear or Almost Clear at Week 12
Description: as for outcome 31
Time Frame: Week 12
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 33.3 | 90.0
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 56.8, 95% CI 2-sided [42.7 to 70.8]

34. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear or Almost Clear at Week 16
Description: as for outcome 31
Time Frame: Week 16
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 31.7 | 91.7
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 59.9, 95% CI 2-sided [46.3 to 73.6]

35. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear or Almost Clear at Week 20
Description: as for outcome 31
Time Frame: Week 20
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 48.3 | 93.3
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 44.9, 95% CI 2-sided [30.8 to 59.1]

36. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear or Almost Clear at Week 24
Description: as for outcome 31
Time Frame: Week 24
Population: ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 38.3 | 93.3
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 55.0, 95% CI 2-sided [41.2 to 68.8]

37. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear at Week 4
Description: as for outcome 31
Time Frame: Week 4
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 0 | 1.7
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p = 0.392, Cochran-Mantel-Haenszel; Adjusted percentage difference = 1.7, 95% CI 2-sided [-2.1 to 5.4]

38. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear at Week 8
Description: as for outcome 31
Time Frame: Week 8
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 1.7 | 10.0
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p = 0.048, Cochran-Mantel-Haenszel; Adjusted percentage difference = 8.4, 95% CI 2-sided [0.1 to 16.7]

39. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear at Week 12
Description: as for outcome 31
Time Frame: Week 12
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 3.3 | 21.7
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p = 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 18.3, 95% CI 2-sided [7.1 to 29.5]

40. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear at Week 16
Description: as for outcome 31
Time Frame: Week 16
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 3.3 | 36.7
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 33.0, 95% CI 2-sided [20.2 to 45.9]

41. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear at Week 20
Description: as for outcome 31
Time Frame: Week 20
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 6.7 | 48.3
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 41.3, 95% CI 2-sided [27.3 to 55.3]

42. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear at Week 24
Description: as for outcome 31
Time Frame: Week 24
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 5.0 | 51.7
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 46.4, 95% CI 2-sided [32.6 to 60.1]

43. Secondary Outcome: Percentage of Participants With Psoriasis Symptoms Scale (PSS) Score of 0 at Week 16
Description: The PSS asks the participant to rate the severity of symptoms of psoriasis in the last 24 hours (pain, redness, itching, and burning) using a 5-point Likert -type scale ranging from 0 (none) to 4 (very severe). The PSS is calculated by summing the scores of the questions and ranges from 0 to 16, where the higher the score, the greater the severity of psoriasis symptoms. NRI was used for missing data.
Time Frame: Week 16
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 5.0 | 25.0
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p = 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 19.8, 95% CI 2-sided [7.6 to 31.9]

44. Secondary Outcome: Percentage of Participants With PSS Score of 0 at Week 24
Description: as for outcome 43
Time Frame: Week 24
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 3.3 | 41.7
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 38.3, 95% CI 2-sided [25.0 to 51.5]

45. Secondary Outcome: PSS Total Score: Change From Baseline to Week 16
Description: The PSS asks the participant to rate the severity of symptoms of psoriasis in the last 24 hours (pain, redness, itching, and burning) using a 5-point Likert -type scale ranging from 0 (none) to 4 (very severe). The PSS is calculated by summing the scores of the questions and ranges from 0 to 16, where the higher the score, the greater the severity of psoriasis symptoms. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 55 | 59
units on a scale | -5.5 (0.52) | -8.7 (0.51)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated by stratified van Elteren test; Test type: Other; p < 0.001, van Elteren test; Least Squares Mean Difference = -3.2, 95% CI 2-sided [-4.5 to -2.0], Standard Error of Mean 0.63

46. Secondary Outcome: PSS Total Score: Change From Baseline to Week 24
Description: as for outcome 45
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 55 | 60
units on a scale | -5.6 (0.49) | -9.5 (0.48)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated by stratified van Elteren test; Test type: Other; p < 0.001, van Elteren test; Least Squares Mean Difference = -3.9, 95% CI 2-sided [-5.1 to -2.7], Standard Error of Mean 0.59

47. Secondary Outcome: Summary of Patient Benefit Index (PBI) at Week 16
Description: The PBI is a patient-reported outcome instrument that assesses the benefit of psoriasis treatment.The PBI assessment consists of 2 steps: before treatment, every participant defines his/her treatment needs according to a standardized list (Patient Needs Questionnaire [PNQ]). After treatment, the participant rates the degree of benefits achieved (Patient Benefits Questionnaire [PBQ]). 25 items are rated on a 5-point scale with values from 0 (not at all) to 4 (very), allowing for "did not apply to me" (5) and missing. For each treatment goal the PNQ importance is derived by dividing the respective PNQ item by the sum of all PNQ items. The weighted sum of each PBQ item with its respective PNQ importance yields the PBI score. An increase in PBI indicates improvement. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 54 | 59
units on a scale | 1.970 (1.1971) | 3.118 (0.8246)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = 1.146, 95% CI 2-sided [0.764 to 1.528]

48. Secondary Outcome: Summary of PBI at Week 24
Description: The PBI is a patient-reported outcome instrument that assesses the benefit of psoriasis treatment. The PBI is a patient-reported outcome instrument that assesses the benefit of psoriasis treatment.The PBI assessment consists of 2 steps: before treatment, every participant defines his/her treatment needs according to a standardized list (PNQ). After treatment, the participant rates the degree of benefits achieved (PBQ). 25 items are rated on a 5-point scale with values from 0 (not at all) to 4 (very), allowing for "did not apply to me" (5) and missing. For each treatment goal the PNQ importance is derived by dividing the respective PNQ item by the sum of all PNQ items. The weighted sum of each PBQ item with its respective PNQ importance yields the PBI score. An increase in PBI indicates improvement. LOCF imputation was used for missing data.
Time Frame: Baseline Week 24
Population: ITT analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 54 | 60
units on a scale | 1.997 (1.2710) | 3.316 (0.7487)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = 1.320, 95% CI 2-sided [0.936 to 1.704]

49. Secondary Outcome: Clinical Severity of Nail Psoriasis (NAPPA-CLIN) Total Score: Change From Baseline to Week 16
Description: The NAPPA-CLIN is an investigator assessment used to assess the severity of nail matrix psoriasis (leukonychia, red spots, dots, nail plate crumbling) and psoriasis of the nail bed (oil drop, splinter haemorrhage, subungual hyperkeratosis, onycholysis). NAPPA-CLIN has been developed from the Nail Psoriasis Severity Index (NAPSI) score, a nail psoriasis-specific score, which in its original version comprises the assessment of matrix and nail bed involvement in every finger and toe by 2 criteria for each nail. The NAPPA-CLIN is a simplified version of the NAPSI which only assesses the least and the worst involved nail of both hands or both feet respectively. Thus, the NAPPA-CLIN scores for hands or feet range from 0 to 16. A higher score indicates a worse involvement. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 56 | 58
units on a scale | -0.4 (0.51) | -2.7 (0.51)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -2.3, 95% CI 2-sided [-3.6 to -1.1], Standard Error of Mean 0.63

50. Secondary Outcome: NAPPA-CLIN Total Score: Change From Baseline to Week 24
Description: The NAPPA-CLIN is an investigator assessment used to assess the severity of nail matrix psoriasis (leukonychia, red spots, dots, nail plate crumbling) and psoriasis of the nail bed (oil drop, splinter haemorrhage, subungual hyperkeratosis, onycholysis). NAPPA-CLIN has been developed from the NAPSI score, a nail psoriasis-specific score, which in its original version comprises the assessment of matrix and nail bed involvement in every finger and toe by 2 criteria for each nail. The NAPPA-CLIN is a simplified version of the NAPSI which only assesses the least and the worst involved nail of both hands or both feet respectively. Thus, the NAPPA-CLIN scores for hands or feet range from 0 to 16. A higher score indicates a worse involvement. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 56 | 58
units on a scale | -0.7 (0.53) | -3.7 (0.54)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-4.3 to -1.6], Standard Error of Mean 0.66

51. Secondary Outcome: Palmoplantar Psoriasis Severity Index (PPASI): Change From Baseline to Week 16
Description: The PPASI is an assessment by the investigator that provides a numeric scoring for psoriasis affecting the hands and feet with scores ranging from 0 to 72. It is a linear combination of percent of surface area of palms and soles that are affected and the severity of erythema, induration, and desquamation. The higher the score, the greater the severity of psoriasis symptoms. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 56 | 60
units on a scale | -0.76 (0.251) | -1.04 (0.249)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p = 0.352, ANCOVA; Least Squares Mean Difference = -0.29, 95% CI 2-sided [-0.90 to 0.32], Standard Error of Mean 0.307

52. Secondary Outcome: PPASI: Change From Baseline to Week 24
Description: as for outcome 51
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 56 | 60
units on a scale | -0.87 (0.242) | -1.17 (0.240)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p = 0.315, ANCOVA; Least Squares Mean Difference = -0.30, 95% CI 2-sided [-0.88 to 0.29], Standard Error of Mean 0.296

53. Secondary Outcome: Body Surface Area (BSA) Affected by Psoriasis: Change From Baseline to Week 4
Description: BSA affected by psoriasis was measured by the physician selecting the participant's right or left hand as the measuring device. For purposes of clinical estimation, the total surface of the palm plus 5 digits was to be assumed to be approximately equivalent to 1% BSA. Measurement of the total area of involvement by the physician was aided by imagining if scattered plaques were moved so that they were next to each other and then estimated the total area involved. A decrease in BSA affected by psoriasis indicates improvement. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 4
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: percentage estimated body surface area
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 58 | 60
percentage estimated body surface area | -0.3 (0.86) | -5.2 (0.86)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -4.8, 95% CI 2-sided [-6.9 to -2.7], Standard Error of Mean 1.06

54. Secondary Outcome: BSA Affected by Psoriasis: Change From Baseline to Week 8
Description: as for outcome 53
Time Frame: Baseline, Week 8
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: percentage estimated body surface area
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 58 | 60
percentage estimated body surface area | -3.5 (1.33) | -12.8 (1.33)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -9.3, 95% CI 2-sided [-12.6 to -6.1], Standard Error of Mean 1.64

55. Secondary Outcome: BSA Affected by Psoriasis: Change From Baseline to Week 12
Description: as for outcome 53
Time Frame: Baseline, Week 12
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: percentage estimated body surface area
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 58 | 60
percentage estimated body surface area | -6.0 (1.22) | -16.2 (1.23)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -10.2, 95% CI 2-sided [-13.2 to -7.2], Standard Error of Mean 1.51

56. Secondary Outcome: BSA Affected by Psoriasis: Change From Baseline to Week 16
Description: as for outcome 53
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: percentage estimated body surface area
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 58 | 60
percentage estimated body surface area | -8.2 (1.22) | -18.0 (1.22)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -9.8, 95% CI 2-sided [-12.8 to -6.8], Standard Error of Mean 1.51

57. Secondary Outcome: BSA Affected by Psoriasis: Change From Baseline to Week 20
Description: as for outcome 53
Time Frame: Baseline, Week 20
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: percentage estimated body surface area
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 58 | 60
percentage estimated body surface area | -9.7 (1.13) | -19.3 (1.13)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -9.6, 95% CI 2-sided [-12.4 to -6.8], Standard Error of Mean 1.39

58. Secondary Outcome: BSA Affected by Psoriasis: Change From Baseline to Week 24
Description: as for outcome 53
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: percentage estimated body surface area
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 58 | 60
percentage estimated body surface area | -9.8 (1.19) | -19.8 (1.19)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -10.0, 95% CI 2-sided [-12.9 to -7.1], Standard Error of Mean 1.47

59. Secondary Outcome: Short Form Health Survey 36, Version 2 (SF-36 V2) Physical Component Summary (PCS) Score: Change From Baseline to Week 16
Description: The SF-36 V2 Health determined participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 comprise the physical component of the SF-36. Scores on each item were summed and averaged (PCS Score; range = 0-100); a positive change from Baseline indicates improvement. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 55 | 59
units on a scale | 2.87 (1.153) | 7.36 (1.135)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p = 0.002, ANCOVA; Least Squares Mean Difference = 4.49, 95% CI 2-sided [1.74 to 7.23], Standard Error of Mean 1.385

60. Secondary Outcome: SF-36 V2 PCS Score: Change From Baseline to Week 24
Description: as for outcome 59
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 55 | 60
units on a scale | 3.68 (1.104) | 8.31 (1.083)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = 4.63, 95% CI 2-sided [2.01 to 7.25], Standard Error of Mean 1.322

61. Secondary Outcome: SF-36 V2 Mental Component Summary (MCS) Score: Change From Baseline: to Week 16
Description: The SF-36 determined participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 5-8 comprise the mental component of the SF-36. Scores on each item were summed and averaged (MCS Score; range = 0-100); a positive change from Baseline indicates improvement. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 55 | 59
units on a scale | 4.20 (1.493) | 10.86 (1.472)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = 6.66, 95% CI 2-sided [3.11 to 10.20], Standard Error of Mean 1.787

62. Secondary Outcome: SF-36 V2 MCS Score: Change From Baseline to Week 24
Description: as for outcome 61
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 55 | 60
units on a scale | 3.56 (1.494) | 11.41 (1.470)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = 7.85, 95% CI 2-sided [4.31 to 11.38], Standard Error of Mean 1.784

63. Secondary Outcome: Patient's Global Assessment (PtGA): Change From Baseline to Week 16
Description: The PtGA is a patient-reported outcome instrument to assess the patient's assessment of disease severity. This self-reported measure is used to assess disease activity using a 4-point scale where a higher score indicates a higher level of disease activity. Disease activity is assessed from 0 ("complete disease control") to 3 ("uncontrolled disease"). LOCF imputation was used for missing data.
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 56 | 59
units on a scale | -1.0 (0.11) | -1.9 (0.11)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-1.2 to -0.7], Standard Error of Mean 0.13

64. Secondary Outcome: PtGA: Change From Baseline to Week 24
Description: as for outcome 63
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 56 | 60
units on a scale | -1.0 (0.11) | -2.0 (0.11)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-1.3 to -0.8], Standard Error of Mean 0.13

65. Secondary Outcome: Hospital Anxiety & Depression Scale (HADS) Total Score-Anxiety: Change From Baseline to Week 16
Description: The HADS was a patient-reported questionnaire used to assess the level of anxiety and depression in the setting of a hospital medical outpatient clinic. The anxiety and depression subscales each have a range from 0-21, higher scores indicated higher levels of anxiety and depression, respectively. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 55 | 59
units on a scale | -2.2 (0.48) | -4.3 (0.47)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.2 to -0.9], Standard Error of Mean 0.57

66. Secondary Outcome: HADS Total Score-Anxiety: Change From Baseline to Week 24
Description: as for outcome 65
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 55 | 60
units on a scale | -1.8 (0.49) | -4.0 (0.48)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -2.3, 95% CI 2-sided [-3.5 to -1.1], Standard Error of Mean 0.59

67. Secondary Outcome: HADS Total Score-Depression: Change From Baseline to Week 16
Description: as for outcome 65
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 55 | 59
units on a scale | -1.8 (0.50) | -4.9 (0.50)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -3.1, 95% CI 2-sided [-4.3 to -1.9], Standard Error of Mean 0.61

68. Secondary Outcome: HADS Total Score-Depression: Change From Baseline to Week 24
Description: as for outcome 65
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 55 | 60
units on a scale | -1.7 (0.54) | -4.8 (0.53)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -3.1, 95% CI 2-sided [-4.4 to -1.8], Standard Error of Mean 0.65

69. Secondary Outcome: Percentage of Participants Achieving Dermatology Life Quality Index (DLQI) Score of 0 or 1 at Week 16
Description: The DLQI is a 10-question questionnaire that asks the participant to evaluate the degree that psoriasis has affected their quality of life in the last week and includes 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment). Responses to each domain are not relevant (0), not at all (0), a little (1), a lot (2), and very much (3). The DLQI is calculated by summing the scores of the questions and ranges from 1 to 30, where 0-1 = no effect on patient's life, 2-5 = small effect, 6-10 = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on patient's life. The higher the score, the more the quality of life is impaired. A 5-point change from baseline is considered a clinically important difference. NRI was used for missing data.
Time Frame: Week 16
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 10.0 | 48.3
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 38.3, 95% CI 2-sided [23.6 to 53.1]

70. Secondary Outcome: Percentage of Participants Achieving DLQI Score of 0 or 1 at Week 24
Description: as for outcome 69
Time Frame: Week 24
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 60 | 60
percentage of participants | 10.0 | 66.7
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-value was calculated from the CMH test adjusted for strata (prior phototherapy [yes/no]); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 56.8, 95% CI 2-sided [42.7 to 70.9]

71. Secondary Outcome: DLQI Total Score: Change From Baseline to Week 16
Description: The DLQI is a 10-question questionnaire that asks the participant to evaluate the degree that psoriasis has affected their quality of life in the last week and includes 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment). Responses to each domain are not relevant (0), not at all (0), a little (1), a lot (2), and very much (3). The DLQI is calculated by summing the scores of the questions and ranges from 1 to 30, where 0-1 = no effect on patient's life, 2-5 = small effect, 6-10 = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on patient's life. The higher the score, the more the quality of life is impaired. A 5-point change from baseline is considered a clinically important difference. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 56 | 59
units on a scale | -9.7 (0.94) | -17.0 (0.94)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with prior phototherapy (yes/no), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -7.4, 95% CI 2-sided [-9.6 to -5.1], Standard Error of Mean 1.15

72. Secondary Outcome: DLQI: Change From Baseline to Week 24
Description: as for outcome 71
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 56 | 60
units on a scale | -11.2 (0.87) | -18.8 (0.87)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -7.6, 95% CI 2-sided [-9.7 to -5.5], Standard Error of Mean 1.06

73. Secondary Outcome: Psoriasis Scalp Severity Index (PSSI): Change From Baseline at Week 16
Description: The physician assessed the severity of scalp psoriasis using the PSSI, which consists of an assessment of erythema, induration, and desquamation on a scale from 0 (none) to 4 (very severe) and the percentage of scalp involved on a scale from 0 (0% of scalp involved) to 6 (90-100% of scalp involved). The composite score is calculated as the sum of symptom scores multiplied by the score for the area of scalp involved. The PSSI ranges from 0 (best) to 72 (worst). A negative change from Baseline indicates improvement. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 56 | 60
units on a scale | -14.6 (1.01) | -21.2 (1.01)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -6.6, 95% CI 2-sided [-9.0 to -4.1], Standard Error of Mean 1.23

74. Secondary Outcome: PSSI: Change From Baseline at Week 24
Description: as for outcome 73
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 56 | 60
units on a scale | -13.9 (1.25) | -22.0 (1.25)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -8.1, 95% CI 2-sided [-11.1 to -5.0], Standard Error of Mean 1.53

75. Secondary Outcome: European Quality of Life 5 Dimensions (EQ-5D-5L) Total Score: Change From Baseline to Week 16
Description: The EQ-5D-5L is a standardized non-disease specific instrument for describing and valuing health-related quality of life. The EQ-5D-5L descriptive system comprises 5 dimensions of health (mobility, self -care, usual activities, pain/discomfort, and anxiety/depression) to describe the subject's current health state. Each dimension comprises 5 levels with corresponding numeric scores, where 1 indicates no problems, and 5 indicates extreme problems. A unique EQ-5D-5L health state is defined by combining the numeric level scores for each of the 5 dimensions and the total score is normalized from -0.594 to 1.000, with higher scores representing a better health state. An increase in the EQ-5D-5L total score indicates improvement. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 55 | 58
units on a scale | 0.083 (0.0179) | 0.171 (0.0176)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = 0.087, 95% CI 2-sided [0.045 to 0.130], Standard Error of Mean 0.0215

76. Secondary Outcome: EQ-5D-5L Total Score: Change From Baseline to Week 24
Description: as for outcome 75
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 55 | 60
units on a scale | 0.106 (0.0155) | 0.165 (0.0152)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p = 0.002, ANCOVA; Least Squares Mean Difference = 0.059, 95% CI 2-sided [0.022 to 0.096], Standard Error of Mean 0.0186

77. Secondary Outcome: EQ-5D-5L Visual Analog Scale (VAS): Change From Baseline to Week 16
Description: The EQ-5D-5L is a standardized non-disease specific instrument for describing and valuing health-related quality of life. The EQ-5D-5L VAS records the participant's self-rated health on a vertical visual analogue scale numbered from 100 (best health imagined) to 0 (worst health imagined). The VAS score from the scale is then entered as a number by the participant. This can be used as a quantitative measure of health outcome that reflects the participant's own judgement. An increase in the EQ-5D-5L VAS score indicates improvement. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 55 | 58
units on a scale | 11.0 (2.32) | 26.0 (2.28)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = 14.9, 95% CI 2-sided [9.4 to 20.5], Standard Error of Mean 2.80

78. Secondary Outcome: EQ-5D-5L VAS: Change From Baseline to Week 24
Description: as for outcome 77
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 55 | 60
units on a scale | 11.6 (2.29) | 28.4 (2.23)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; P-values were calculated using ANCOVA with strata (phototherapy [yes/no]), baseline value, and treatment in the model; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = 16.8, 95% CI 2-sided [11.4 to 22.2], Standard Error of Mean 2.73

79. Secondary Outcome: Nail Psoriasis Severity Index (NAPSI): Change From Baseline to Week 16
Description: The NAPSI score is calculated by summing the scores of all the nails which for each nail are the sum of the nail matrix score and nail bed score. Each of these is scored as 0=none, 1=present in 1/4 nail, 2=present in 2/4 nail, 3=present in 3/4 nail, 4=present in 4/4 nail. Each nail has a matrix score (0-4) and a nail bed score (0-4). The total nail score is the sum of those 2 (nail matrix and nail bed) individual scores (0-8). The sum of the total score of all involved fingernails is then the total NAPSI score. The NAPSI score is calculated only if all questions in the case report form are completed. A negative change from Baseline indicates improvement. LOCF imputation was used for missing data.
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 56 | 58
units on a scale | -2.2 (2.13) | -13.6 (2.14)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; [analysis description as in outcome 25, analysis 1]; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -11.4, 95% CI 2-sided [-16.6 to -6.2], Standard Error of Mean 2.64

80. Secondary Outcome: NAPSI: Change From Baseline to Week 24
Description: as for outcome 79
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 56 | 58
units on a scale | -4.4 (2.18) | -18.1 (2.19)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; [analysis description as in outcome 25, analysis 1]; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -13.7, 95% CI 2-sided [-19.1 to -8.4], Standard Error of Mean 2.70

81. Secondary Outcome: Participants With Baseline NAPSI ˃0: Change From Baseline to Week 16
Description: as for outcome 79
Time Frame: Baseline, Week 16
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 33 | 42
units on a scale | -4.2 (3.11) | -21.4 (2.86)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; [analysis description as in outcome 25, analysis 1]; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -17.3, 95% CI 2-sided [-24.8 to -9.8], Standard Error of Mean 3.75

82. Secondary Outcome: Participants With Baseline NAPSI ˃0: Change From Baseline to Week 24
Description: as for outcome 79
Time Frame: Baseline, Week 24
Population: ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fumaderm | Risankizumab
Number analyzed (Participants) | 33 | 42
units on a scale | -6.0 (3.03) | -27.5 (2.79)
Statistical Analysis 1: Comparison: Fumaderm vs Risankizumab; [analysis description as in outcome 25, analysis 1]; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -21.5, 95% CI 2-sided [-28.8 to -14.2], Standard Error of Mean 3.66

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 15 weeks after the last dose of risankizumab (up to 31 weeks) or until 1 week after the last dose of Fumaderm(R) (up to 25 weeks).
Description: Safety analysis set included all participants enrolled in the study and who received at least 1 dose of study drug (N = 117).
Arm/Group | Fumaderm | Risankizumab
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/60
Serious Adverse Events (participants affected / at risk) | 2/57 | 1/60
Other Adverse Events (participants affected / at risk) | 54/57 | 45/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fumaderm (N=57) | Risankizumab (N=60)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fumaderm (N=57) | Risankizumab (N=60)
Lymphopenia (Blood and lymphatic system disorders) | 8 (9) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 11 (13) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 26 (34) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 32 (57) | 4 (4)
Nausea (Gastrointestinal disorders) | 9 (12) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (4)
Bronchitis (Infections and infestations) | 3 (3) | 3 (3)
Influenza (Infections and infestations) | 3 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 26 (32) | 35 (47)
Rhinitis (Infections and infestations) | 3 (4) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 7 (15) | 5 (6)
Migraine (Nervous system disorders) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (8) | 2 (2)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Flushing (Vascular disorders) | 23 (28) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT03255382/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT03255382/SAP_001.pdf